CLINICAL TRIAL: NCT06917066
Title: Spanish Prospective Registry: MYval Induced Late and EArly Conduction Disturbances (MYLEAD)
Brief Title: MYLEAD Spanish Prospective Registry
Acronym: MYLEAD
Status: Recruiting | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Collaborators: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Principal Investigator, Ignacio J. Amat Santos, Coordinator of Interventional Cardiology Unit, Hospital Clínico Universitario de Valladolid
Other Study IDs: PS-24-22-C
Record Dates: First submitted 2025-03-13; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Severe Aortic Valve Stenosis
Keywords: Severe Aortic Valve Stenosis; TAVR; Myval Transcatheter Heart Valve
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Severe Aortic Valve Stenosis: All patients with Severe Aortic Valve Stenosis undergoing TAVR using Myval Transcatheter Heart Valve
  Interventions: Procedure: TAVR

INTERVENTIONS:
Procedure: TAVR — TAVR procedure using Myval Transcatheter Heart Valve

SUMMARY:
Investigator-initiated, prospective, multicentre registry, whose objectives are: 1/ to evaluate the incidence of conduction defects and the need of pacemaker implantation post-procedure, at discharge, at 30 days and at 1 year post Myval transcatheter heart valve deployment, and 2/ To evaluate the factors determining in-hospital and late (at 30 days and 1 year) conduction defects post Myval transcatheter heart valve.

Patients with Severe Aortic stenosis undergoing TAVR using Myval Transcatheter Heart Valve that meet all inclusion criteria and any exclusion criteria will be able to participate in this study if they sign the informed consent. Electrocardiogram, echocardiogram and computed tomography will be performed to patients at different time points (Baseline, post-procedure, discharge, 30 days and 1 year post procedure) and their parameters will be added into a dedicated REDCAP database.

DETAILED DESCRIPTION:
Study Design: Investigator-initiated, prospective, multicentre registry. Study Phase: Phase IV.

Study Objectives:

1. To evaluate the incidence of conduction defects and the need of pacemaker implantation post-procedure, at discharge, at 30 days and at 1 year post Myval transcatheter heart valve deployment.
2. To evaluate the factors determining in-hospital and late (at 30 days and 1 year) conduction defects post Myval transcatheter heart valve.

Description of the study protocol:

* Patients meeting the inclusion and exclusion criteria will be enrolled after taking informed consent. The baseline data and electrocardiogram (ECG), echocardiogram and computed tomography parameters will be added into a dedicated REDCAP database.
* TAVR will be performed as per the standard procedure using Myval Transcatheter Heart Valve.
* The ECG parameters post procedure, at discharge, at 30 days and at 1 year post-procedure will be noted using the REDCAP database.
* Based on these ECG parameters, analysis will be done to look for mean variations of PR and QRS segments, atrio-ventricular block, bundle branch block or need for pacemaker from baseline to post-procedure, at discharge, at 30 days and at 1 year post procedure.
* Echocardiogram parameters at 30 days (optional) and at 1 year post procedure will be noted using the REDCAP database.
* Statistical analysis will be done using IBM SPSS Statistics and R software.

Study duration:

* Inclusion stage: Patients will be recruited during the index procedure; if the patient meets all the inclusion criteria and any exclusion criteria and accepts to participate. ECG, echocardiogram and computed tomography will be done at baseline and the relevant information will be entered into the electronic database.
* In-hospital stage: Postprocedural and predischarge ECGs will be obtained and all the required clinical information will be gathered before discharge.
* Follow up stage: Clinical follow-up will be performed at 30 days and at 1 year post procedure, and the required ECG parameters will be obtained. At the 30-day follow-up, echocardiographic variables will be collected if the centers are available to perform echocardiograms or if an echocardiogram has been performed to the patients for other reasons within the determined period. In the 1-year follow-up, echocardiographic variables collected by clinical practice will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years of age)
* Patients with Severe Aortic stenosis undergoing TAVR using Myval Transcatheter Heart Valve.

Exclusion Criteria:

* Patients with pre-existing permanent pacemaker.
* Patients unable or unwilling to follow up for pre and post procedure clinical assessments and investigations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with of Severe Aortic stenosis undergoing TAVR using Myval Transcatheter Heart Valve who meet all inclusion criteria and any exclusion criteria in 32 centers in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of rhythm disorders | 30 days
  Presence of any of the following conduction defects detected in 12-lead ECG:
  1. Atrial Fibrillation
  2. Pacemarker
  3. Left bundle branch block
  4. Right bundle branch block
  6) 1st degree AVB 7) Other conduction disturbances

SECONDARY OUTCOMES:
Presence of rhythm disorders | Postprocedural, 7 days, 1 year
  Presence of any of the following conduction defects detected in 12-lead ECG:
  1. Atrial Fibrillation
  2. Pacemarker
  3. Left bundle branch block
  4. Right bundle branch block
  6) 1st degree AVB 7) Other conduction disturbances
Duration of PR interval | Postprocedural, 7 days, 30 days, 1 year
  Duration of PR interval (ms) measured in ECG
Duration of QRS complex | Postprocedural, 7 days, 30 days, 1 year
  Duration of QRS complex (ms) measured in ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No